CLINICAL TRIAL: NCT06934174
Title: Cultural Adaptation of a Web-Based App (myPlan Thailand) to Empower and Support Friends and Family of Intimate Partner Violence Survivors
Acronym: IPV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boromarajonani College of Nursing, Khon Kaen (Other)
Collaborators: Johns Hopkins University (Other); Auckland University of Technology (Other); Notre Dame of Maryland University (Unknown); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Tipparat Udmuangpia, Assistant Professor, Boromarajonani College of Nursing, Khon Kaen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BoromarajonaniCNKK; 5K43TW012296 (NIH)
Record Dates: First submitted 2025-04-10; First posted 2025-04-18 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Intimate Partner Violence (IPV); Social Support; Empowerment; mHealth; Effectiveness
Keywords: Intimate partner violence; Friends/Family memeber; Safety; Social support; mHealth intervention; Thailand
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WeSafe (myPlan Thailand: Friends and Family) (Experimental): WeSafe, a Web-Based App (myPlan Thailand) is a culturally tailored web-based app designed to empower and support friends and family of IPV survivors. It gathers key data on survivors' demographics, relationship status, living situation, and children's ages to personalize the safety support plan. The app delivers comprehensive IPV information through text, videos, images, and illustrations, addressing culturally specific issues. It guides users in setting priorities through pairwise comparisons and includes a risk assessment tool adapted from Danger Assessment (DA)-Thailand. Based on the inputs, myPlan Thailand provides a tailored plan with supportive strategies, communication scripts, advocacy tips, self-care resources, and child safety strategies, enhancing overall safety and well-being.
  Interventions: Behavioral: WeSafe (myPlan Thailand: Friends and Family); Behavioral: DV learning
- DV learning (Active Comparator): Control group. The control condition will be the publicly-available Thai-language DV learning launched in 2019.49 This app screens users for Domestic violence (physical, psychological, and sexual violence), and provides information about 6 modules include 1. Understanding situation of domestic violence 2. Key principles of helping survivors 3. Guideline for helping survivors 4. Case management and working with multi professionals 5. Legal Proceedings and Justice System Processes for Domestic Violence and Intimate Partner Violence Cases 6. Selfcare for providers. This platform put the knowledge from understanding the basic situation through practical intervention for providers and other people who are interested in. It is optional to get the certificate if participants have 80% pass rate on quizzes.
  Interventions: Behavioral: WeSafe (myPlan Thailand: Friends and Family); Behavioral: DV learning

INTERVENTIONS:
Behavioral: WeSafe (myPlan Thailand: Friends and Family) — WeSafe, a Web-Based App (myPlan Thailand) is a culturally tailored web-based app designed to empower and support friends and family of IPV survivors. It gathers key data on survivors' demographics, relationship status, living situation, and children's ages to personalize the safety support plan. The app delivers comprehensive IPV information through text, videos, images, and illustrations, addressing culturally specific issues. It guides users in setting priorities through pairwise comparisons and includes a risk assessment tool adapted from Danger Assessment (DA)-Thailand. Based on the inputs, myPlan Thailand provides a tailored plan with supportive strategies, communication scripts, advocacy tips, self-care resources, and child safety strategies, enhancing overall safety and well-being.
Behavioral: DV learning — Control group. The control condition will be the publicly-available Thai-language DV learning launched in 2019.49 This app screens users for Domestic violence (physical, psychological, and sexual violence), and provides information about 6 modules include 1. Understanding situation of domestic violence 2. Key principles of helping survivors 3. Guideline for helping survivors 4. Case management and working with multi professionals 5. Legal Proceedings and Justice System Processes for Domestic Violence and Intimate Partner Violence Cases 6. Selfcare for providers. This platform put the knowledge from understanding the basic situation through practical intervention for providers and other people who are interested in. It is optional to get the certificate if participants have 80% pass rate on quizzes.

SUMMARY:
This research will support and empower friends/family (F/F) of intimate partner violence (IPV) survivors in Thailand, where IPV is critical and common, and survivors first and foremost seek help for abuse from their F/F. myPlan app (www.myPlanapp.org) is a free mobile evidence-based intervention app to prevent IPV. The app was first developed in the United States (US) and has been disseminated to high-income countries (e.g., New Zealand, Canada, Australia) and lowincome (Kenya). One new hope for improving survivors' psychological and well-being is adapting and introducing the myPlan app for the concerned friends/family who support survivors in Thailand.

Therefore, the propose of this longitudinal research study, Cultural Adaptation of a Web-Based App (myPlan Thailand) to Empower and Support Friends/Family of Intimate Partner Violence Survivors in Thailand, will have two consecutive phases with three aims: 1) To tailor the myPlan app content for concerned F/F members of Thai IPV survivors, 2) To integrate the adapted myPlan app content for concerned F/F members of Thai IPV survivors, 3) To test the feasibility and acceptability of the adapted myPlan app with concerned F/F members of Thai IPV survivors. Phase 1 (Year 1-2) will achieve aim 1-2 to tailor the myPlan app with Thai survivors and friends/family. The investigators will review current content and conduct in-depth interviews with survivors and concerned F/F members on social norms associated with IPV, informal support systems and the role/responsibility in helping survivors, safety strategies used by concerned F/F members and negative consequences for both survivor and F/F member providing support. Moreover, in phase 1, the adapted content will be pilot tested with concerned F/F members of survivors by using cognitive techniques and theater-testing methodology.

Phase 2 (Year 3-4) will achieve aim 3 to test the feasibility and acceptability of the adapted myPlan app with F/F. The investigators will conduct a two-group RCT design with concerned F/F member randomized to receive a) the myPlan app for F/F member, or b) standard usual-care safety planning information. Primary outcomes for F/F members include change in knowledge and attitudes towards IPV and F/F empowerment to plan and take safety support survivor. Secondary outcomes will examine change in F/F' distress, frustration and consequences for supporting the survivor. This phase will also collect feasibility and acceptability data to informed a planned R01 submission in Year 3 of the study. The K43 application outlines a four-year plan to support a candidate who is a nursing instructor with 15 years of work in diverse projects, settings, and disciplines; which positions her for a successful career as an independent researcher in research field of intimate partner violence. The career development plan provides a sequence of carefully selected training and mentoring experiences, including coursework to increase research capacity, leadership skills, mentored research leading to a R01 proposal, peer reviewed publications, and professional networking, that will catapult this research to the next level of research achievement. The team will be a collaboration between the Boromarajonani College of Nursing Khon Kaen (BCNKK), Khon Kaen One Stop Crisis Center (OSCC), Johns Hopkins University (JHU), Notre Dame of Maryland University (NDM), and Auckland University of Technology (AUT), New Zealand.

ELIGIBILITY:
Inclusion Criteria:

* being female or males who have a female friend currently (past 6 months) experiencing IPV
* Thai speaking/reading
* At least 18 years old
* Have access to a safe smart-phone or computer with internet
* Have safe email address
* Living in Thailand

Exclusion Criteria:

* Cannot speak/reading Thai
* Less than age 18 years old
* Cannot access to a safe smartphone or computer with internet
* Not living in Thailand

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Knowledge and Attitudes towards IPV | Baseline, 1 month, 3 months, and 6 months
  Knowledge and attitudes toward IPV measurement will be adapted from the Inventory of Beliefs about Intimate Partner Violence (IBIPV) with a 22-item self-report scale, with a seven-point response scale designed to assess participants' explicit attitudes toward IPV, and from the literature around friends/family response as describe by survivors and engagement behavior. There are 22 items, group into three subscales.The Justifying Partner Violence subscale (JPV; six items; e.g., "Sometimes abuse of the woman helps resolve conflictsbetween partners") deals with general behaviours of victims and abusers which may be used to legitimise or justify IPV.The Victims Responsible for Violence subscale (VRV; nineitems; e.g., "Battered women are responsible for battering,because they provoke it") deals with victim behaviours whichmay lead to women being blamed for IPV. Finally, theAbuser Responsible for Violence subscale (ARV; sevenitems; e. g., "Abusers are responsible for batterin
Empowerment to plan and take actions to safely support survivor | Baseline, 1 month, 3 months, and 6 months
  Empowerment to plan and take actions to safely support survivor will be measured by the Personal Progress Scale-Revised, which is a 28 items, 7-point Likert scale with focus on the important role of resilience and personal empowerment for women. The scale includes item such as "I want to help other women like me improve the quality of their lives). The reliability coefficient for this scale is .85.
The Supportive Behaviors checklist | Baseline, 1 month, 3 months, and 6 months
  This tool is a 23-item self-report scale designed to assess supportive actions undertaken by friends or family when concerned about a loved one's abusive relationship. Participants indicate for each item whether, in the past six months, they engaged in specific supportive behaviors and rate if they were helpful using a three-point response scale ("No (1)," "Yes(2), but I didn't think it was helpful," "Yes(3), and I thought it was helpful"). Items cover a range of actions-from active listening and validating concerns to facilitating safety measures and connecting with professional resources-providing an evaluative insight into both behavioral engagement and perceived effectiveness in supporting IPV survivors.

SECONDARY OUTCOMES:
Distress, frustration, and negative consequences for supporting the survivors | Baseline, 1 month, 3 months, and 6 months
  stress, frustration, and negative consequences for supporting the survivors (e.g., anger by friend/ family member) will assess the decisional conflict immediately post intervention. It will be adapted from the Decisional Conflict Scale (DCS) with 12 items test whether using the myPlan app to helps a friends/family to understand the advantages/ disadvantages of options for helping their friends in an abusive relationship, and to know her values related to those options (e.g., "I know my options for helping my friend who is in an unhealthy.", I am clear about which reasons for helping my friend are most important to me.", "I have enough advice to make decisions about helping my friend who is in an unhealthy relationship." The scale is a Likert scale; 5 = strongly agree;...1 = strongly disagree.
Feasibility and Acceptability | 6 months
  The feasibility and acceptability measurement will be guided by the Weiner et al (2017). 12 items for acceptability (e.g. number of times participated signed on, use of content in each section, barriers/facilitators of use) and 8 items for measuring feasibility (study procedures, recruitment/retention rates, time to recruit participant target, rate of completion of intervention). The score will be a 5-point Likert scale; 5 = strongly agree;....1= strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Tipparat Udmuangpia, PhD,MS,RN, Principal Investigator — Boromarajonani College of Nursing, Khon Kaen
Locations (1):
- Maliwan Thaewbao, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No